CLINICAL TRIAL: NCT04481867
Title: Patient Perception and Radiographic Assessment of Sinus Lifting Procedure Using Densah Bur Versus Ostetome . A Randomized Clinical Trial
Brief Title: Patient Perception and Radiographic Assessment of Sinus Lifting Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Amr Heshmat, lecturer od prosthodontic dep,, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sinus lift densah bur
Record Dates: First submitted 2020-07-13; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Dental Implant Failed
Keywords: Sinus lifting; CBCT

STUDY DESIGN:
Intervention Model Description: randomized control trail
Who Masked: Outcomes Assessor
Masking Description: blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm :densah bur group (Active Comparator): at the maxillary molar area for implant placement ,,just after making initial drilling perforation close to the sinus floor, the direction of the drill is reversed and the cutting speed is raised to 1200 rpm, then 2 successive densah burs are used to elevate sinus membrane 2 mm and to prepare implant hole to the selected implant size .for both groups the selected implant size, 4.2 mm width and 10 mm. length
  Interventions: Procedure: densah bur
- control group :osteotome group (Other): at the maxillary molar area for implant placement .a set of concave osteotomes with different dimensions sequentially used to widen the osteotomy site by surgical mallet. Osteotome 2.5 mm is inserted into the osteotomy firstly to a depth of 1 mm away from the sinus floor with light malleting by the nylon cap mallet then 3 mm osteotome is used to fracture up the sinus floor and finally 3.5 mm osteotome is tapped gently to elevate the sinus floor to the desired depth of the implant in the maxillary sinus.
  Interventions: Procedure: densah bur

INTERVENTIONS:
Procedure: densah bur — osseodensification densah bur

SUMMARY:
This study aimed to evaluate the clinical complications that might be presented with osteotome and densah burs, as well as to assess the new bone generated at 6 months post-operatively using CBCT. The study hypothesis was that densah bur would show comparable results to osteotome-mediated sinus lifting

DETAILED DESCRIPTION:
Maxillary posterior edentulous area rehabilitation with implants is usually not an easy procedure and is considered a challenge to many prosthodontists. This is due to pneumatization of the maxillary sinus, poor bone density and volume, and difficult accessibility of this area. After tooth loss, the maxillary sinus tends to enlarge into the remaining residual ridge because of poor bone density and lack of functional stimulation by teeth.1 Rehabilitation with dental implants in the maxillary posterior area depends on the quantity and quality of bone available for implant placement. In order to place the implant in the best prosthetic position, regenerative surgical techniques are usually essential to correct the initial anatomical situation.2 Summer in 1994 introduced a less invasive technique than the lateral approach for sinus floor elevation, called the closed sinus lifting. Summer classified it in to osteotome sinus floor elevation and bone added osteotome sinus floor elevation. Osteotome depends on condensing the bone in implant bed site and pushing it laterally and upward, which raises the sinus floor. Although being successful and non-invasive, Summer's technique showed several surgical problems as heat generation-induced necrosis if not well irrigated, and delayed implant secondary stability, as well as some patient-related drawbacks as headache and vertigo.3 Fortunately, in 2014 Salah Huwais introduced new burs called densah burs that help preservation of bone health by condensing bone rather than removing it. Accordingly, this process was labeled osseodensification. In the past few years since the introduction of densah burs, limited number of studies evaluated its efficiency as well as patient perception to the procedure. 4 It is well established that cone beam computed tomography (CBCT) gives more profound and accurate assessment of pre- and post-operative implant sites. However, a meta-analysis was published in 2018 showed that most previous studies on lifting procedures used conventional 2D techniques, and very few applied CBCT as the diagnostic modality. This heterogeneity highly affected the quality of evidence retrieved. 5 This study aimed to validate the clinical complications that might be presented with osteotome and densah burs, as well as to assess the new bone generated at 6 months post-operatively using CBCT. The study hypothesis was that densah bur would show comparable results to osteotome-mediated sinus lifting.

ELIGIBILITY:
Inclusion Criteria:

* the residual bone height at the site of implant placement was 8 mm or less. All patients were in a good health, non-smokers with no systemic, immunologic or debilitating diseases that could affect normal bone healing. Their edentulous ridges were covered with optimal thickness of mucoperiosteum with no signs of inflammation, ulceration or scar tissue and sufficient inter arch space was adequate for future prosthesis

Exclusion Criteria:

* smokers bad oral hygiene systemic disease

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Clinical patient perception | 7 days postoperative
  assessment with Health-Related Quality of Life (HRQOL) questionnaire

SECONDARY OUTCOMES:
Radio-graphic (CBCT) assessment | preoperative and 6 month postoperative
  New bone length around the implant ,in millimetre

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Heshmat, lecturer, Study Director — faculty of dentistry ,Cairo Uni
Locations (1):
- Faculty of dentistry ,Cairo Uni, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Result] Almutairi AS, Walid MA, Alkhodary MA. The effect of osseodensification and different thread designs on the dental implant primary stability. F1000Res. 2018 Dec 5;7:1898. doi: 10.12688/f1000research.17292.1. eCollection 2018. PMID 31131085
- [Result] Padhye NM, Padhye AM, Bhatavadekar NB. Osseodensification -- A systematic review and qualitative analysis of published literature. J Oral Biol Craniofac Res. 2020 Jan-Mar;10(1):375-380. doi: 10.1016/j.jobcr.2019.10.002. Epub 2019 Nov 2. PMID 31737477